CLINICAL TRIAL: NCT00779649
Title: MoviPrep® Versus HalfLytely® for Colon Cleansing: An Investigator-blinded, Randomized Trial.
Brief Title: MoviPrep® Versus HalfLytely®, Low-VolUme PEG Solutions for Colon Cleansing: An InvesTigator-blindEd, Randomized, Trial
Acronym: LUSTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Associates of New York, LLP (Other)
Responsible Party: Lawrence B Cohen, MD, Research Associates of New York
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: LUSTER
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Colonoscopy
Keywords: Colonoscopy,; Prep; MoviPrep; HalfLytely; The effectiveness of colonoscopy preps
MeSH Terms: interventions — Bisacodyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MoviPrep (Active Comparator)
  Interventions: Other: MoviPrep Kit
- HalfLytely (Active Comparator)
  Interventions: Other: HalfLytely and Bisacodyl Tablets Bowel Prep Kit

INTERVENTIONS:
Other: MoviPrep Kit — Diet: At noon the day prior to the procedure, patients will begin a clear liquid diet. Patient will discontinue any ingestion by mouth 4 hours prior to the procedure.
  Purgative: Starting at 6pm the evening before the procedure, patient will ingest 250 ml of MoviPrep® at 15 minute intervals until 1 liter is consumed. Following this, an additional 500 ml (approximately 16 oz) of clear liquids will be consumed. The next day, 6 hours before the procedure, the patient will repeat ingestion of one liter MoviPrep® over the course of an hour, again ingesting 250 ml at 15 minute intervals. Patient will then ingest an additional 500 ml (approximately 16 oz) of clear liquid following the MoviPrep® consumption.
  Arms: MoviPrep
Other: HalfLytely and Bisacodyl Tablets Bowel Prep Kit — Diet: Patients will refrain from solid food and have only clear liquids starting 8 am on the day before colonoscopy. In addition, patients will consume nothing by mouth, except clear liquids, from the time the preparation is completed until midnight. Patients will be instructed not to eat or drink anything from midnight until after the colonoscopy is completed.
  Purgative: At noon on the day prior to colonoscopy patients will swallow (not chew or crush) 2 bisacodyl delayed release tablets (10 mg). Once the initial bowel movement has occurred (1 - 6 hours after taking the bisacodyl tablets), or if there has been no bowel movement, not more than 6 hours after ingestion of the bisacodyl tablets patients will then drink the reconstituted HalfLytely® solution over 1 hour and 20 minutes. Patients will drink one 8-oz glass every 10 minutes until the two liters is completed
  Arms: HalfLytely

SUMMARY:
A properly prepared colon is vital to the success of any colonoscopy. The purpose of this study is to determine which colon prep, MoviPrep or HalfLytely is the superior prepping agent.

DETAILED DESCRIPTION:
To demonstrate, by direct visualization, the superior overall colon cleansing efficacy of MoviPrep®, to that of HalfLytely® and Bisacodyl Tablets Bowel Prep Kit in adults undergoing colonoscopy

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent.
2. Is scheduled for colonoscopy within 30 days of screening
3. Is a male or non-pregnant, non-lactating female, at least 18 years of age and not greater than 75 years of age. Females of childbearing potential must be using an acceptable form of birth control
4. Is able to communicate effectively with study personnel.

Exclusion Criteria:

1. Known allergy or hypersensitivity to any constituent of MoviPrep® (polyethylene glycol, sodium sulfate, sodium chloride, potassium chloride, sodium ascorbate, ascorbic acid), or any constituent of HalfLytely with bisacodyl (lactose (anhydrous), NF, microcrystalline cellulose NF, croscarmellose sodium NF, magnesium stearate NF, eudragit L 30-55, talc USP, gelatin, calcium sulfate (anhydrous) NF, confections sugar, kaolin USP, sucrose NF, opalus pink, beeswax, carnuba wax, saccharine.
2. Use of any drugs that may affect GI motility such as laxatives, stool softeners, promotility agents, products to prevent diarrhea, purgatives and enemas during the study. Non-systematically absorbed medications (e.g. milk of magnesia, MiralaxTM) can be held for 24 hours prior to taking the study medication. Systematically absorbed medications can be held based upon their half-life and length of activity.
3. History of renal insufficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study will be a comparison of mean overall colon cleansing scores for each treatment arm, determined by the ratings on the Physician Questionnaire. | one year from the trial start date

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence B Cohen, MD, Principal Investigator — New York Gastroenterology Associates, L.L.P